CLINICAL TRIAL: NCT02529241
Title: An Open-label, Single Dose, Parallel Design, Phase I Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Oral Dosage Form of LCB01-0371 in Healthy Volunteers
Brief Title: An Open-label, Single Dose, Parallel Design, Phase 1 Clinical Study of LCB01-0371
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCB01-0371-15-1-01
Record Dates: First submitted 2015-08-12; First posted 2015-08-20 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: LCB01-0371 (Experimental): Period 1: LCB01-0371 Tablet 400 mg Period 2: LCB01-0371 Tablet 400 mg
  Interventions: Drug: Group 1:LCB01-0371; Drug: Group 2:LCB01-0371
- Group 2: LCB01-0371 (Experimental): Period 1: LCB01-0371 Tablet 800 mg Period 2: LCB01-0371 Tablet 1200 mg
  Interventions: Drug: Group 1:LCB01-0371; Drug: Group 2:LCB01-0371

INTERVENTIONS:
Drug: Group 1:LCB01-0371 — 1. Period:LCB01-0371 Tablet 400 mg
  2. Period: LCB01-0371 Tablet 400 mg
Drug: Group 2:LCB01-0371 — 1. Period:LCB01-0371 Tablet 800 mg
  2. Period: LCB01-0371 Tablet 1200 mg

SUMMARY:
To investigate pharmacokinetics, safety and tolerability of LCB01-0371, LCB01-0371-B after a single oral dose in healthy male subjects.

To investigate safety, tolerability of LCB01-0371 after a single oral dose in healthy male subjects.

DETAILED DESCRIPTION:
An Open-label, Single dose, Parallel design, Phase I Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Oral dosage form of LCB01-0371 in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male between 20 and 40 years of age at the time of screening
2. Agree to continue to use a medically reliable dual contraception and not to donate sperm in this protocol for the duration of the study and for 28 days after last dose of investigational product
3. Capable of giving written informed consent, willing to participate in this clinical trial, and willing to comply with all study requirements

Exclusion Criteria:

1. History of gastrointestinal problem (e.g. Crohn's disease, gastro-intestinal ulcer) within 6 months possibly affecting absorption of clinical trial drugs, or history of surgery (except simple appendectomy and herniotomy)
2. History of hypersensitivity reaction or history of clinically significant hypersensitivity reaction to LCB01-0371 or same class of the study drugs (linezolid) or other drugs including aspirin and antibiotics
3. History of clinically significant disease such as allergic or anaphylactic reaction to drug, cardiovascular, peripheral vascular system, skin, mucous membrane, eye, otorhinolaryngologic system, respiratory, musculoskeletal, infection disease, Gastrointestinal system , liver, biliary system, endocrine, kidney, urogenital system, nervous system, psychiatric system, blood dyscrasia, tumor, fracture, problem(s)
4. blood donation and transfusion within 60 days prior to screening visit
5. Treatment with an other investigational product or Participation in other bioequivalence test within 90 days prior to screening visit
6. Use medication which expected to influence in this study within 30 days prior to screening visit
7. smokers over 10 cigarettes per day within 30 days prior to screening visit or unable to stop smoking in this protocol for the duration of the study from first dose of investigational product
8. drinkers over 3 glasses alcohol drink per week within 30 days prior to screening visit or unable to stop drinking in this protocol for the duration of the study from first dose of investigational product
9. positive result at urine drug screening test or urine nicotine test at screening visit
10. positive result at serum test(hepatitis B, hepatitis C, HIV, syphilis) at screening visit
11. corrected QT interval >450 msec or significant abnormalities on screening ECG
12. other: Patients considered unable perform for the study by the investigator concerning

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Peak Plasma Concentration (Cmax) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours
Pharmacokinetics: time to maximum concentration (Tmax) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours

SECONDARY OUTCOMES:
Number of Adverse Event | participants will be followed after hospital stay, an expected average of 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea